CLINICAL TRIAL: NCT05890898
Title: Virtual Reality: An Interventional Study Comparing the Use of Virtual Reality to Nitrous Oxide for Analgesia During Dental Procedures on Pediatric Patients
Brief Title: Virtual Reality vs Nitrous Oxide in Pediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1000
Record Dates: First submitted 2023-05-03; First posted 2023-06-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Dentistry
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Nitrous Oxide, then Virtual Reality Goggles (Experimental): Control group will receive the standard of care dental treatment with under nitrous sedation (N2O) and will have a second visit where Virtual Reality(VR) goggles will be used instead of N2O.
  Interventions: Behavioral: Virtual Reality Headset; Drug: Nitrous Oxide
- Treatment: Virtual Reality Goggles, then Nitrous Oxide (Experimental): The treatment group will receive the standard of care dental treatment with VR googles first and will have a second visit under N2O will be used instead of VR.
  Interventions: Behavioral: Virtual Reality Headset; Drug: Nitrous Oxide

INTERVENTIONS:
Behavioral: Virtual Reality Headset — To determine if virtual reality headsets can reduce a patients pain level instead of using the standard Nitrous. This may provide a alternate to patients who cannot receive nitrous if pain or anxiety can be reduced effectively.
Drug: Nitrous Oxide — Nitrous Oxide is the current standard of care being used and will be compared to the use of the VR headsets.

SUMMARY:
Two groups of pediatric patients between the ages of 4 to 12 years old will be examined in this study. Control group will receive the standard of care dental treatment with under nitrous sedation (N2O) and will have a second visit where Virtual Reality(VR) goggles will be used instead of N2O. The treatment group will receive the standard of care dental treatment with VR googles first and will have a second visit where N2O will be used instead of VR. Procedures performed in all groups will be restorative treatments, which can include intraoral anesthetic injections, placing dental fillings, crowns, and the extractions of teeth. In group 1, A specific VR headset, the "Oculus Quest 2" will be used. Through the headset, a video will be played for the child during a dental procedure.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled, interventional therapy utilizing virtual reality goggles as a method of distraction. Data will be collected during and after the procedure on the type of behavior displayed and the child's response to standardized questions. Pediatric patients aged 4-12 years who only require nitrous sedation to complete painful dental treatment which necessitates anesthesia will be included in this study. These patients exhibit Frankl 2-3 behavior, requiring behavior guidance in order to complete the procedure. Frankl 1 or 4 children, those who do not need behavior guidance at all, or children with heavy behavior guidance who would not be able to complete the procedure, will be excluded.

Participants will be recruited in the clinic, during a new patient exam, routine hygiene or operative dentistry appointment. Following the Frankl behavior score diagnosis, an evaluation of behavior will happen during the beginning of the appointment, specifically watching for acceptance of treatment plan, openness to conversation, and any defiant behaviors or crying.

The parent and child being recruited for the study will be informed of the nature of the study, the possible risks benefit and alternatives, and written consent will be obtained from the parent or legal guardian. Assent from child 7 to 12 will also be required as well. The qualifying patient will enter the operatory and be admitted into the study. Participants will be briefed on how the study will proceed, and will be randomized into a control group or treatment group. The groups will be selected at random prior to treatment in the study. Both Groups will use of Faces, Legs, Arms, Crying Consolability(FLACC) Scale, WongBaker FACES, and Houpt Behavior scales to access the pain or discomfort of subjects. Patients will rate their pain using the Wong-Baker FACES Pain Scale by indicating which face best depicts the pain they are experiencing. Each face has a corresponding number: 0 = doesn't hurt at all to 10 = hurts as much as you can imagine. Patients will be observed during injection and assessed by the operator using the Faces, Legs, Arms, Crying Consolability (FLACC) scale. Each category will be rated from 0 to 2. Zero indicating normal positions and no sign of discomfort and 2 indicating discomfort in movements or unable to console/comfort. Patients will be observed during the procedure using the Houpt Behavioral Scale. Each category is scored on the 0-2 scale which results in a total score of 0-10. Assessment of Behavioral Score: 0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 = Moderate pain, 7-10 = Severe discomfort/pain.

Patients receiving N2O during their visit will follow the standard of care procedures. The VR goggles will be placed on the head and in front of the eyes. Patients using the goggles are automatically set to start media as soon as the wearer dons them. The patient will be reclined, and placed in an ideal setting, and the goggles will be calibrated to the patient's current view. The dental procedure will then follow. Most procedures require a local anesthetic injection, and if the patient receives this injection, participants will be graded with FLACC score during the injection. At the end of the procedure the child will be evaluated using the Wong-Baker FACES scale, the Houpt Crying and Movement Scales, and a survey will be given to the patient to be completed.

Participants will participate in the study during two restorative dental appointments, however, some patients may need more than two visits. Participants who require multiple restorative treatments will only being include in the study during first two visits and no other research activities will occur after. Most appointments are projected to last a maximum of 1 hour. The limiting factor in all treatment in this study, will be the participant's willingness to participate in future appointments.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric dental patients age 4-12 years
* Require two restorative procedures that includes injection of anesthesia
* American Society of Anesthesiologists (ASA) physical status classification 1 or 2

Exclusion Criteria:

* Have health issues that prevent use of VR Oculus headset,
* Hypersensitivity to audio-visual devices that can lead to seizures
* ASA physical status classification 3 or 4

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Rate of effectiveness virtual reality goggles reduce pain | 12 months
  To determine whether the use of distraction via virtual reality headset can be as effective as nitrous oxide for purposes of anxiolysis and analgesia during dental treatment. The FLACC scale will be used to help measure this outcome.
  Patients will be observed during injection and assessed by the operator using the Faces, Legs, Arms, Crying Consolability (FLACC) scale. Each category will be rated from 0 to 2. Zero indicating normal positions and no sign of discomfort and 2 indicating discomfort in movements or unable to console/comfort.
Rate of effectiveness virtual reality goggles reduce pain | 12 months
  To determine whether the use of distraction via virtual reality headset can be as effective as nitrous oxide for purposes of anxiolysis and analgesia during dental treatment. The WongBaker scale will be used to help measure this outcome.
  Patients will rate their pain using the Wong-Baker FACES Pain Scale by indicating which face best depicts the pain they are experiencing. Each face has a corresponding number: 0 = doesn't hurt at all to 10 = hurts as much as you can imagine.

SECONDARY OUTCOMES:
Rate of effectiveness of virtual reality distraction to nitrous oxide | 12 months
  To determine if there is a difference in the effectiveness between the use of the standard nitrous oxide and VR distraction. The Houpt scales will be used to help measure this outcome.
  Patients will be observed during the procedure using the Houpt Behavioral Scale. Each category is scored on the 0-2 scale which results in a total score of 0-10. Assessment of Behavioral Score: 0 = Relaxed and comfortable, 1-3 = Mild discomfort, 4-6 = Moderate pain, 7-10 = Severe discomfort/pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger, Danville, Pennsylvania, United States